CLINICAL TRIAL: NCT04870268
Title: A Tailored Step-up Approach for Moderate to Critical Acute Pancreatitis in the Late Phase: a Cohort Study
Brief Title: Late Phase Acute Pancreatitis: a Tailored Step-up Approach
Acronym: TSA
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Simone guadagni, Principal Investigator, University of Pisa
Other Study IDs: example-1
Record Dates: First submitted 2021-04-13; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Acute Pancreatitis
Keywords: acute pancreatitis; walled-off necrosis; surgical treatment; quality of life
MeSH Terms: conditions — Pancreatitis | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 22 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PD group: percutaneous drainage group
  Interventions: Procedure: percutaneous drainage
- END group: endoscopic approach group
  Interventions: Procedure: endoscopic approach
- INT group: surgical internal derivation of WON group
  Interventions: Procedure: surgical internal derivation of WON
- NE group: surgical necrosectomy group
  Interventions: Procedure: surgical necrosectomy

INTERVENTIONS:
Procedure: percutaneous drainage
  Groups: PD group
Procedure: endoscopic approach
  Groups: END group
Procedure: surgical internal derivation of WON
  Groups: INT group
Procedure: surgical necrosectomy
  Groups: NE group

SUMMARY:
Several interventional and surgical procedures are available to treat moderate-to-critical acute pancreatitis (AP) in its late phase. The ongoing debate on these options, together with the scarcity of reported mid-term follow-up information in the Literature, prompted the investigators to conduct a review of our surgical experience, focused on those issues. The investigators reviewed retrospectively all the patients treated for moderate-to-critical AP according to Determinant-Based Classification (DBC), in the last nine years. Patients treated conservatively or operated within 4 weeks of the onset of the pancreatitis were excluded. All the included patients were managed following a "tailored" step-up approach, and divided into four groups, according to the first interventional procedure performed: percutaneous drainage (PD), endoscopic approach (END), internal derivation (INT), and necrosectomy (NE). In-hospital and mid-term follow-up variables, including a quality-of-life assessment, were analyzed and compared.

DETAILED DESCRIPTION:
The following variables were evaluated: sex, age, severity of inflammation according to the DBC classification, PA etiology, CT scan severity index according to Balthazar criteria , clinical prognostic score using bedside index of severity of acute pancreatitis (BISAP) score.

Total length of hospitalization, operative management, necrosis cultures, total and post-interventional Intensive Unit Care (ICU) were also recorded and analyzed together with the in-hospital morbidity, mortality and re-admissions.

Patients were checked after discharge within 14 days and followed monthly as outpatients by gastroenterologists. A CT scan was performed within 4 months, or before in case of recurrent symptoms. During the follow-up, the English Standard Short Form 36 (SF-36) questionnaire was used to evaluate the general quality of life at three and six months, one and two years. The SF-36 examines 8 areas consisting of social and physical function, physical and emotional well-being, bodily pain, vitality, mental health and overall general health perception. At the six-month follow-up, the patients also completed a specific questionnaire about the pancreatic function. In particular, the total score takes in consideration abdominal pain using visual analogue pain score, diarrhea, unintentional weight loss, new onset of diabetes and use of enzyme supplementation. The score ranges between zero to five (all symptoms present). The work has been reported in line with the STROCSS criteria

ELIGIBILITY:
Inclusion Criteria:

* patients treated at our referral Center for moderate to critical AP, as classified by Determinant-Based Classification of Acute Pancreatitis Severity

Exclusion Criteria:

* patients who had undergone conservative treatment,
* patients who has been operated within 4 weeks (early phase)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The cohort sample was divided into four groups, according to the first type of the interventional or surgical management performed
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2012-01; Primary Completion 2020-04 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Satisfaction assessed by the SF-36 (36-Item Short Form Survey) | 1 year
  English Standard Short Form 36 (SF-36) questionnaire is used to evaluate the general quality of life. The SF-36 examines 8 areas consisting of social and physical function, physical and emotional well-being, bodily pain, vitality, mental health and overall general health perception. The eight scaled scores are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Candio G, Guadagni S, Furbetta N, Gianardi D, Palmeri M, Di Franco G, Bianchini M, Gambaccini D, Marciano E, Cervelli R, Marchi S, Morelli L. A "tailored" interventional and surgical management for moderate to critical acute pancreatitis in late phase: a cohort study. Langenbecks Arch Surg. 2022 Nov;407(7):2833-2841. doi: 10.1007/s00423-022-02557-x. Epub 2022 May 31. PMID 35639137

DOCUMENTS (1):
  • Study Protocol (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/68/NCT04870268/Prot_000.pdf